CLINICAL TRIAL: NCT02608294
Title: Influence of Kinesio Taping® in Paretic Tibialis Anterior Muscle at Joint Dynamics During Patient Gait and Balance After Stroke: A Pilot Study
Brief Title: Influence of Kinesio Taping® in Paretic Tibialis Anterior Muscle During Patient Gait and Balance After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Danielly Laís Pereira Lima Gomes, Degree in Physiotherapy, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15238913.9.0000.5208
Record Dates: First submitted 2015-11-15; First posted 2015-11-18 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Stroke
Keywords: stroke; gait; balance
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Group (Experimental): Kinesio Taping Procedure application with 35% strain.
  Interventions: Device: Kinesio Taping
- Sham Group (Sham Comparator): Kinesio Taping Sham procedure application without strain.
  Interventions: Device: Kinesio Taping Sham

INTERVENTIONS:
Device: Kinesio Taping — The patient is placed on a stretcher, his ankle positioned in plantar flexion and inversion, a measure was held between Point A and B with a tape measure, right after the KT was removed from the paper and cut to the same extent. The KT was pulled to its maximum limit and measured with a tape for a second evaluator. This measure found after the maximum tensile strain represented 100% and a rule of three was applied in order to find the 35% voltage for muscle activation. After finding the measure of 35% strain in centimeters, the evaluator cut KT this measurement and the same was discarded. Finally the tape was positioned at Point A; pulled up to Point B; and fixed. This procedure was carried out with the ankle positioned in plantar flexion and inversion.
  Arms: Experimental Group
Device: Kinesio Taping Sham — The sham group received the tape applied without tension. The patient was positioned supine; the ankle was placed in a neutral position (90 degrees); and measured between Point A and Point B with a tape measure placed on the skin was performed. Once registered this measure in centimeters the evaluator cut the KT with the same measure, but without the presence of paper attached to it to ensure that there was no tension, because the KT needs a minimum voltage to be applied on paper. After measured and cut the KT, it was applied to the patient in the supine position with the ankle positioned at 90 degrees with no traction.
  Arms: Sham Group

SUMMARY:
A pilot study was conducted, randomized, triple-blind study with allocation concealment. Which consisted in the application of KT in the anterior tibial muscle for 24 hours. 14 subjects were randomized into 2 groups: intervention (with voltage) and sham (no pressure). Patient's gait footage was shot in the opening balance of phases, average balance and initial contact (first without the application of Kinesio Taping and after 24 hours of application) to be measured the angles of the ankle joints, knee and hip. Balance was assessed by the Biodex Balance System platform, configured to analyze the postural stability in level eight. The mean differences were assessed (MD) between groups and confidence interval (CI) of 95%.

DETAILED DESCRIPTION:
The sample was selected from the list of patients waiting for care in Kinesiology Laboratory and Functional Assessment of the Department of Physical Therapy, Federal University of Pernambuco - UFPE where the operation was performed. In the period from May to July 2014. The study was approved by the Ethics Committee in Research with Human beings of the Health Sciences Center of UFPE, CAAE 15238913.9.0000.5208. On admission, patients were informed about the research, met the free and informed consent. Randomization was taken by randomization.com site, and the allocation concealment was done with opaque and sealed envelopes.

Procedures for application of Kinesio Taping As for the protocol, the intervention group and the sham group underwent the same way care for skin preparation. Trichotomy, when necessary was held; the skin was cleaned with alcohol and dry with a paper towel.

They were used as a reference point between the proximal fibular head and the tibial tuberosity (point A) and the apex of the first metatarsal (Point B). The experimental group received the voltage for activating muscle and were positioned to receive the application of KT in accordance with the manual taping kinesio - Kenzo Kase method. And only one tape mark was used, which is recommended by the Kinesio Taping Association.

KT application in the intervention group The patient was placed on a stretcher in the supine position, his ankle was positioned in plantar flexion and inversion (maximum amplitude achieved passively by the patient), a measure was held between Point A and B with a tape measure, then immediately KT was removed from the paper and cut to the same extent. The KT was pulled to its maximum limit and measured with a tape for a second evaluator. This measure found after the maximum tensile strain represented 100% and a rule of three was applied in order to find the 35% voltage for muscle activation. The tension of KT was calculated to ensure an approximate voltage to all participants in the intervention group.

After finding the measure of 35% strain in centimeters, the evaluator cut KT this measurement and the same was discarded. Finally the tape was positioned at Point A; pulled up to Point B; and fixed. This procedure was carried out with the ankle positioned in plantar flexion and inversion, maximum amplitude achieved passively by the patient.

KT application in the sham group The sham group received the tape applied without tension. The patient was positioned supine; the ankle was placed in a neutral position (90 degrees); and measured between Point A and Point B with a tape measure placed on the skin was performed. Once registered this measure in centimeters the evaluator cut the KT with the same measure, but without the presence of paper attached to it to ensure that there was no tension, because the KT needs a minimum voltage to be applied on paper. After measured and cut the KT, it was applied to the patient in the supine position with the ankle positioned at 90 degrees with no traction.

Images of funding for procedures The patient was markers (pressure ball) in the lower limbs at predetermined anatomical points: head of the fifth metatarsal, below the midpoint of the lateral malleolus, head of the fibula, lateral femoral condyle and greater trochanter of the femur. They recorded images with a Digital Camcorder (CANON PowerShot A2600) fixed to a tripod. Environmental calibration was performed by a board calibration with 120 cm high, with a tag of 60 cm, which was calibrated at the midpoint of the focus of the camcorder.

During recording were filmed right and left profiles of the patient. This was dressed in shorts containing a side screen, allowing viewing and palpation of anatomical points already mentioned.

After receiving the markers at the anatomical points the patient was encouraged to walk on a flat track with eight meters long by three times, the two central meters used. The 1ºgravação was carried out without application of KT and the patient was instructed to walk at their normal pace of the march. After application of KT patient returned and was released after 24 hours. They were placed markers in pre-determined anatomical points and the patient was encouraged to walk again on track in its normal rhythm of the march to the 2nd recording taking place with the same conditions of the first day.

1. Balance evaluation The tool used to assess postural balance was the Biodex Balance System, a device used in order to check and / or train in closed kinetic chain static and dynamic postural stability in patients with one foot or bipedal. The apparatus consists of two components: an adjustable platform 12 different levels of stability, being "1" the more unstable level and "12" as static level and a display, which is given a feedback of the location of the center of mass of the individual. The level used in Postural Stability test was 8 (following the manual protocol) for providing low loss of balance and postural adjustment the patient uses the ankle strategy, in which there is greater participation of the gastrocnemius muscles to a previous imbalance and tibialis anterior for a subsequent imbalance.

The display demonstrates a point on the screen as center of pressure of the patient and their displacement is attributed to the balance of the body that is quantified by CP movement in the anterior / posterior direction (generating the index of anterior / posterior stability: IAP) and medial / side (generating medial stability index / side: IML) together IAP and the IML result in the general stability index (GSE), the higher the value the higher indices the body of the swing, ie, the greater the instability in patients. In addition to providing the percentage of evaluation time within each zone (A, B, C and D) and each quadrant (I, II, III and IV).

The assessment of the balance through the BBS used the level 8 in the test Postural Stability. The test was performed three times with a duration of 20 seconds, with 10 seconds interval between repetitions, with the first evaluation, four replications and excluding the first to reduce the potential effects of learning. The result was considered a final average of three tests for each variable. All values are saved on your computer and recorded in a spreadsheet by the evaluator.

To carry out the balancing test, age and the patient's height were recorded on the equipment, then the participant was asked rise in the BBS platform and the positioning of the feet was also recorded. Was asked to what patient adopt a comfortable posture with arms along the body, did not move the feet of the place throughout the test, put the ball in the center of the picture and look at the phone's display throughout the duration of the evaluation .

Satisfaction Rating Twenty-four hours after application of patients returned to service and KT was removed. Then the patients were asked about their satisfaction with the use of Kinesio with the question: "Did you notice positive differences regarding the use of KT to facilitate the walk? ". For the answer patients had two options "yes" or "no." And they could express verbally how and where was this positive difference.

Analysis of the images The images were captured in the sagittal plane in video form and then transferred to a computer and analyzed by the Free Software Tracker - Tool analysis and physical modeling videos. The software was used to analyze joint angles of knee, hip and ankle. They were selected frames of three gait phases: opening balance, average balance and initial contact. At each stage of it was marked angles of the ankle, knee and hip; each angle was measured 3 times to produce an average angular. The image calibration done in software using a tag in the center of the track in black with 60 cm length.

Statistical analysis Data were tabulated in Microsoft Office Excel 2007 and then reviewed by a researcher blinded to the status of the groups. Statistical analysis was performed using SPSS 13.0 for Windows versions. To characterize the sample was used descriptive analysis using measures of central tendency (mean) and dispersion (standard deviation) for quantitative variables and frequency for categorical variables. Due to the small sample size, non-parametric tests were used. For intergroup analysis was performed Mann-Whitney test and intra-group analysis was done Wilcoxon obtaining differences between the groups and their respective confidence intervals (95% CI). The level of significance with statistical difference was p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stroke Ischemic or Hemorrhagic proven by clinical examination and imaging;
* Stroke with minimal evolution of six months (chronic hemiparetic more than 6 months after injury);
* Kinetic-functional Diagnostic hemiparesis, spasticity degrees with between 1 and 2 in Ashworth scale modified for muscle group of ankle plantar flexor;
* People over 21 years;
* What do not use assistive devices while driving;
* Absence of cognitive impairment (Mini-Mental State Examination MMSE - illiterate ≤ 15 points, 1-11 years of schooling ≤ 22 with higher education to 11 years ≤ 27)

Exclusion Criteria:

* Presented range of motion to lowest passive dorsiflexion than 5 degrees;
* If there were missing during the intervention period;
* Presented clinical comorbidities that interfere in the intervention such as high blood pressure or cardiac arrhythmias
* And submit pathological deformities of the lower limbs or presence of scabs on malleolus

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-07; Primary Completion 2014-09 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Ankle angle during 1 gait cycle | 30 seconds
  Angle measured from the ankle joint during some phases of the gait cycle.

SECONDARY OUTCOMES:
Balance | 20 seconds
  Observation of the patient's balance on the balance measurement platform (Biodex Balance System).

CONTACTS AND LOCATIONS:
Overall Officials: Danielly Gomes, B.S., Principal Investigator — Universidade Federal de Pernambuco
Locations (1):
- Departamento de Fisioterapia - Universidade Federal de Pernambuco, Recife, Pernambuco, Brazil

REFERENCES:
- [Background] Mostafavifar M, Wertz J, Borchers J. A systematic review of the effectiveness of kinesio taping for musculoskeletal injury. Phys Sportsmed. 2012 Nov;40(4):33-40. doi: 10.3810/psm.2012.11.1986. PMID 23306413
- [Background] Williams S, Whatman C, Hume PA, Sheerin K. Kinesio taping in treatment and prevention of sports injuries: a meta-analysis of the evidence for its effectiveness. Sports Med. 2012 Feb 1;42(2):153-64. doi: 10.2165/11594960-000000000-00000. PMID 22124445